CLINICAL TRIAL: NCT03667170
Title: Study of KN035 as Monotherapy in Patients With Advanced Mismatched Repair Deficient (dMMR) or Microsatellite Instability-High (MSI-H) Solid Tumors
Brief Title: KN035 for dMMR/MSI-H Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-CN-006
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor
Keywords: MSI-H; dMMR; Colorectal cancer; Non-Colorectal Cancers
MeSH Terms: conditions — Colorectal Neoplasms | interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with MSI-H/dMMR (Experimental): patients receive 600 mg of the KN035 Subcutaneously every 3 weeks
  Interventions: Biological: KN035

INTERVENTIONS:
Biological: KN035 — subcutaneous injection

SUMMARY:
In this study, patients with previously-treated locally-advanced or metastatic mismatched repair deficient (dMMR) or microsatellite instability-high (MSI-H) colorectal carcinoma (CRC) and other solid tumors will be treated with KN035 monotherapy.

For colorectal cancer participants, who are required to have been previously treated with standard therapies , other solid tumor participants, who are required to have been previously treated with at least one line of systemic standard of care therapy.

DETAILED DESCRIPTION:
Later-line therapies after failure of standard treatments for advanced colorectal and non-colorectal cancer patients are limited. Mismatch repair (MMR) deficiency or microsatellite instability-high (MSI-H) played a role of positive predictive factor, which had been documented after the pembrolizumab and nivolumab trial were reported, for PD-1 blockade monotherapy in patients with advanced colorectal and non-colorectal cancers.

In this study, patients with previously-treated locally-advanced or metastatic mismatched repair deficient (dMMR) or microsatellite instability-high (MSI-H) colorectal carcinoma (CRC) and other solid tumors will be treated with KN035 monotherapy.

For colorectal cancer participants, who are required to have been previously treated with standard therapies. For other solid tumor participants, who are required to have been previously treated with at least one line of systemic standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic colorectal carcinoma or other malignant solid tumors.
* Confirmed MMR deficient or MSI-H status.
* At least one measureable lesion.
* Eastern Cooperative Oncology Group performance status of 0 or 1 .
* Life expectancy of greater than 12 weeks.
* Adequate hematologic and organ function.

Exclusion Criteria:

* Currently participated in a study of an investigational agent and received trial treatment, or used an investigational device within 4 weeks of the first dose of medication in this study. Patients who have had specific anti-tumor treatment within 2 weeks prior to the first dose of study.
* Patients who have not recovered to CTCAE Grade 1 or better from related side effects of any prior antineoplastic therapy.
* Has received prior therapy with an immune check point agonist/inhibitor.
* Patients who have undergone major surgery within 4 weeks of dosing of investigational agent.
* Has a known additional malignancy that is progressing or requires active treatment within the past 5 years.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment.
* Patients who have known history of infection with HIV.
* Patients with evidence of interstitial lung disease.
* Patients who have known history of any major cardiac abnormalities.
* Patient who is not willing to apply highly effective contraception during the study.
* Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  per Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST 1.1) assessed by central imaging vendor

SECONDARY OUTCOMES:
ORR | Up to approximately 2 years
  per Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST 1.1) assessed by investigator
Disease Control Rate (DCR) | Up to approximately 2 years
  per RECIST 1.1 assessed by central imaging vendor and investigator
Duration of Response (DOR) | Up to approximately 2 years
  per RECIST 1.1 assessed by central imaging vendor and investigator
Progression-Free Survival (PFS) | Up to approximately 2 years
  per RECIST 1.1 assessed by central imaging vedor and investigator
Overall Survival (OS) | Up to approximately 2 years
  Calculated by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking Universtiy Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui C, Wang J, Wang C, Xu T, Qin L, Xiao S, Gong J, Song L, Liu D. Model-informed drug development of envafolimab, a subcutaneously injectable PD-L1 antibody, in patients with advanced solid tumors. Oncologist. 2024 Sep 6;29(9):e1189-e1200. doi: 10.1093/oncolo/oyae102. PMID 38982653
- [Derived] Li J, Deng Y, Zhang W, Zhou AP, Guo W, Yang J, Yuan Y, Zhu L, Qin S, Xiang S, Lu H, Gong J, Xu T, Liu D, Shen L. Subcutaneous envafolimab monotherapy in patients with advanced defective mismatch repair/microsatellite instability high solid tumors. J Hematol Oncol. 2021 Jun 21;14(1):95. doi: 10.1186/s13045-021-01095-1. PMID 34154614